CLINICAL TRIAL: NCT06414148
Title: A Phase II Open-Label, Multi-Centre Study of Minimal Residual Disease-Directed Consolidation With Epcoritamab or Epcoritamab-Lenalidomide-Rituximab Post Anti-CD19 CAR TCell Therapy for Large B-Cell Lymphoma (EpLCART)
Brief Title: MRD-Directed Consolidation With Epcor-only or Epcor-R2 Post Anti-CD19 CAR TCell Therapy for Large B-Cell Lymphoma
Acronym: EpLCART
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/012
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Relapsed/Refractory Large B-cell Lymphoma
Keywords: Minimal Residual Disease; Large B-Cell Lymphoma; Anti-CD19; CAR T; ctDNA; Lymphoma; DLBCL; HGBL; Epcoritamab; Lenalidomide; Rituximab
MeSH Terms: conditions — Recurrence; Neoplasm, Residual; Lymphoma | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Intervention Model Description: A phase II open-label, two-arm randomised non-comparative, multicentre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): EPCORITAMAB (EPCOR-ONLY)
  Interventions: Drug: Epcoritamab
- Arm B (Experimental): EPCORITAMAB, LENALIDOMIDE AND RITUXIMAB (EPCOR-R2)
  Interventions: Drug: Epcoritamab, lenalidomide and rituximab

INTERVENTIONS:
Drug: Epcoritamab — Epcoritamab will be administered as a 28-day cycle. In Cycle 1 and 2, epcoritamab will be given with step up dosing in Cycle 1. From Cycle 3 onwards dosing will be on Day 1 and 15 of each cycle.
  Arms: Arm A
Drug: Epcoritamab, lenalidomide and rituximab — Treatment with epcoritamab will be administered following the same dosing schedule as Arm A. On days where rituximab and/or lenalidomide are also due, epcoritamab should be administered last.
  Patients will receive lenalidomide once daily on Day 1-21 of each 28-day cycle, starting at Cycle 1 through to Cycle 6.
  Patients will receive rituximab administered by intravenous (IV) infusion on Day 1, 8, 15 and 22 of Cycle 1 and on Day 1 only of Cycles 2-6.
  Arms: Arm B

SUMMARY:
This is a Phase II open-label, two-arm randomised non-comparative, multi-centre study to evaluate the efficacy of Epcor-only (Epcoritamab alone) or Epcor-R2 (Epcoritamab, lenalidomide and rituximab) as consolidation post anti-CD19 CAR T-cell therapy for patients that have responded by conventional criteria but who are at high risk of progression by virtue of being Minimal Residual Disease (MRD) positive as determined by a Circulating Tumour DNA (ctDNA) assay.

DETAILED DESCRIPTION:
Patients who have received CAR T-cell therapy for Relapsed/Refractory Large B-Cell Lymphoma, are in Complete Metabolic Response (CMR) or Partial Metabolic Response (PMR) and MRD positive post CAR T-cell infusion are potentially eligible. Once these patients have provided their consent, they will enter the screening phase. All events of Cytokine Release Syndrome (CRS), Haemophagocytic Lymphohistiocytosis (HLH)/Macrophage Activation Syndrome (MAS), Immune-Effector Cell Associated Neurologic Syndrome (ICANS), or infection must have completely resolved. Additionally, patients must have adequate organ and haematological function, and an ECOG performance status of up to 2.

Patients deemed eligible for the study will be randomised to receive Epcor-only (Arm A) or Epcor-R2 (Arm B) for 6 cycles. The primary endpoint is CMR by Lugano 2014 criteria at month 12 post CAR T-cell infusion.

Patients will undergo an interim response assessment after 2 cycles of treatment. Patients that complete the full 6 cycles of treatment or that discontinue treatment for any reason will have an End of Treatment visit and a Safety Follow-up visit at 60 days after Day 1 of Cycle 6. Patients with non-Progressive Disease (PD) then enter the follow-up phase of the study where they will undergo response assessments at month 12, 15, 18 and 24 after CAR T-cell infusion. Patients with PD at any time will complete a Progression visit. Patients that have completed the month 24 Follow-up visit or that they have progressed will be followed for survival and new anti-lymphoma therapy only. All patients will be followed for 2 years after the last patient randomised received the CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 16 years old at the time of signing the patient information and consent form (PICF)
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
3. A diagnosis of relapsed/refractory large B-cell lymphoma
4. Received Therapeutic Good Administration (TGA) approved anti-CD19 CAR T-cell therapy as the most recent large B-cell lymphoma treatment.
5. Partial metabolic response (PMR) or complete metabolic response (CMR) as per the Lugano criteria on the most recent PET/CT performed at any point between Day +25 and Day +100 post CAR T-cell infusion, when compared with the most recent PET/CT prior to CAR T-cell infusion.
6. MRD positive by a ctDNA assay on a blood sample taken at any point between Day +25 and Day +100 post CAR T-cell infusion.
7. Adequate haematological function documented within 7 days prior to randomisation
8. Adequate cardiac function.
9. Adequate renal function, documented within 7 days prior to randomisation
10. Adequate hepatic function documented within 7 days prior to randomisation
11. Complete resolution of cytokine release syndrome (CRS), macrophage-activation syndrome (MAS)/haemophagocytic lymphohistiocytosis (HLH) or immune effector cell-associated neurotoxicity syndrome (ICANS) related to prior CAR T-cell therapy.
12. Female patients of childbearing potential (FCBP) must be willing to follow the contraceptive method/procedure as outline in the PICF
13. Sexually active males must agree to use a condom during sexual contact with a pregnant female or a FCBP for the course of the study through to 4 months after the last dose of epcoritamab, even if he has undergone a successful vasectomy
14. Women must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction. Men must also not donate sperm during the trial and for 4 months after receiving the last dose of epcoritamab
15. The patient understands the purpose of the trial and procedures required for the trial which includes compliance with the protocol requirements and restrictions listed in the PICF and in this protocol

Exclusion Criteria

1. A history of Grade 4 CRS or ICANS related to prior CAR T-cell therapy
2. Patients whose lymphoma is known to be CD20 negative on the most recent biopsy prior to CAR T-cell therapy
3. Ongoing active bacterial, viral, fungal, mycobacterial, parasitic, or other infection requiring systemic treatment
4. Progression or relapse within 3 months after a regimen containing a bispecific antibody targeting CD3 and CD20
5. A diagnosis of primary central nervous system (CNS) lymphoma
6. Active secondary CNS involvement of lymphoma at time of screening
7. A known history or current autoimmune disease or other diseases resulting in permanent immunosuppression
8. Known cognitive impairment would place the patient at increased risk of complications from ICANS
9. A known history of hepatitis B serology consistent with acute or chronic infection
10. A known history of hepatitis C serology consistent with acute or chronic infection
11. A known history of testing positive for human immunodeficiency virus (HIV)
12. Any comorbidity conferring a life expectancy of < 5 years (e.g., second malignancy) or that in the opinion of the site investigator may significantly impact the ability to complete the trial therapy and follow-up or affect the interpretation of results
13. Exposed to live or live attenuated vaccine within 4 weeks prior to signing the PICF.
14. Women who are pregnant or lactating
15. Known hypersensitivity to epcoritamab, lenalidomide, rituximab, tocilizumab or their excipients
16. Presence of any psychological, social or geographical or other condition for which participation would not be in the best interest of the patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Epcor-only (epcoritamab alone) or Epcor-R2 (epcoritamab, lenalidomide and rituximab) consolidation as assessed by conventional (Lugano 2014) response criteria at month 12 after the CART infusion | From start of treatment till the end of study, assessed up to approximately 12 months

SECONDARY OUTCOMES:
To evaluate the safety of time-limited Epcor-only or Epcor-R2 consolidation post CAR T-cell therapy according to number of participants with treatment-related adverse events (AE) as assessed by CTCAE v5.0 | From start of treatment till the end of study, assessed up to approximately 48 months
The efficacy as assessed by molecular and conventional response criteria at defined time points with Event Free Survival (EFS) analyses | From start of treatment till the end of study, assessed up to approximately 48 months
The efficacy as assessed by molecular and conventional response criteria at defined time points with Overall Survival (OS) analyses | From start of treatment till the end of study, assessed up to approximately 48 months
The deliverability as assessed by rates of completion of the course of therapy | From start of treatment till the end of study, assessed up to approximately 6 months
The deliverability as assessed by protocol-defined number of dose-reductions of lenalidomide | From start of treatment till the end of study, assessed up to approximately 6 months

OTHER OUTCOMES:
Correlation between tumour/immunological associations (using cytokine/chemokine profiles, clonal kinetics and phenotypic changes) and response (EFS and OS) | From start of treatment till the end of study, assessed up to approximately 48 months
Correlation between tumour/immunological associations (using cytokine/chemokine profiles, clonal kinetics and phenotypic changes) and treatment toxicity (number of participants with treatment-related AE) | From start of treatment till the end of study, assessed up to approximately 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, MBBS, D Med Sc, FRACP, FRCPA, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Alfred Hospital, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No